CLINICAL TRIAL: NCT05797142
Title: The Effect of Virtual Reality-Based Relaxation Program on Pain Intensity, Anxiety Level and Patient Satisfaction in Patients to be Applied With Endoscopy
Brief Title: Virtual Reality-Based Relaxation Program on Pain Intensity, Anxiety Level in Patients to be Applied With Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Sabahattin Zaim University (Other)
Responsible Party: Principal Investigator, Zülfünaz ÖZER, Principal Investigator, Istanbul Sabahattin Zaim University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020-11
Record Dates: First submitted 2023-03-10; First posted 2023-04-04 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Anxiety; Pain
Keywords: virtual reality glasses; Pain; Anxiety; Endoscopy
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This study is an experimental study with pre-test and post-test control groups
Who Masked: Participant
Masking Description: Virtual reality glasses and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- : Virtual reality glasses (Experimental): Beginning 1-2 minute before the start of the procedure, the patients will be watched (30 minutes) with an android mobile phone inserted into the Cardboard Super Flex Binoculars Glasses, with a music background, licensed product "Secret Garden", during the procedure (30 minutes).
  Interventions: Other: Virtual reality glasses
- Control group (No Intervention): Routine maintenance will be applied

INTERVENTIONS:
Other: Virtual reality glasses — Beginning 1-2 minute before the start of the procedure, the patients will be watched (30 minutes) with an android mobile phone inserted into the Cardboard Super Flex Binoculars Glasses, with a music background, licensed product "Secret Garden", during the procedure (30 minutes).
  Arms: : Virtual reality glasses

SUMMARY:
This study was conducted to evaluate the effect of relaxation exercise with VR (Virtual Reality) glasses on pain severity, anxiety level, physiological symptoms of anxiety and satisfaction in patients undergoing endoscopy.

DETAILED DESCRIPTION:
Beginning 1-2 minute before the start of the procedure, the patients will be watched (30 minutes) with an android mobile phone inserted into the Cardboard Super Flex Binoculars Glasses.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Ability to communicate adequately
* Absence of psychiatric problems
* Volunteering to participate in the research

Exclusion Criteria:

Those who have communication problems

* Those with psychiatric problems
* Being unconscious

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-07-08 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | Baseline (Before endoscopy)
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.
Visual Analog Scale | 5 minute after endoscopy
  The patients were asked to mark their level of pain during relaxation or activities on a 10 cm vertical or horizontal line. In addition, there were forms which were numbered from 1-10 or from 1-100. The number 0 is found at the beginning of the line, and the number 10 is located at the end of the line. A value of 0 shows that there is no pain, and the value 10 expresses unendurable pain. GAS is a common scale in the assessment of pain level. A patient is asked to mark the perceived pain on this line, and the marked point is measured in cm.

SECONDARY OUTCOMES:
Anxiety Assessment Scale | Baseline (Before endoscopy)
  Patients will be asked to show their anxiety levels before and after the procedure on a 10 cm long horizontal line. Anxiety Assessment Scale, line has 0 at the beginning and 10 at the end. 10 means very extreme anxiety and 0 means no anxiety.
Anxiety Assessment Scale | 5 minute after endoscopy
  Patients will be asked to show their anxiety levels before and after the procedure on a 10 cm long horizontal line. Anxiety Assessment Scale, line has 0 at the beginning and 10 at the end. 10 means very extreme anxiety and 0 means no anxiety.
Physiological Symptoms of Anxiety Follow-up Form | Baseline (Before endoscopy)
  This form was created by the researcher to record blood pressure, heart rate, respiratory rate and peripheral oxygen saturation (SpO2) value.
Physiological Symptoms of Anxiety Follow-up Form | 1 minute after endoscopy
  This form was created by the researcher to record blood pressure, heart rate, respiratory rate and peripheral oxygen saturation (SpO2) value.
Virtual Reality Glasses Application Satisfaction Form | 5 minute after endoscopy
  In this form, there are questions prepared in line with the relevant literature in order to determine the satisfaction with the video watched with virtual reality glasses.

CONTACTS AND LOCATIONS:
Overall Officials: Zülfünaz Özer, PhD, Principal Investigator — Istanbul Sabahattin Zaim University
Locations (1):
- Istanbul Sabahattin Zaim University, Faculty of Health Sciences, Istanbul, Turkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Genc H, Korkmaz M, Akkurt A. The Effect of Virtual Reality Glasses and Stress Balls on Pain and Vital Findings During Transrectal Prostate Biopsy: A Randomized Controlled Trial. J Perianesth Nurs. 2022 Jun;37(3):344-350. doi: 10.1016/j.jopan.2021.09.006. Epub 2022 Apr 7. PMID 35397973